CLINICAL TRIAL: NCT05023551
Title: A Phase 1 Study of DSP-0390 in Patients With Recurrent High-Grade Glioma
Brief Title: Study of DSP-0390 in Patients With Recurrent High-Grade Glioma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSP-0390-101
Record Dates: First submitted 2021-07-27; First posted 2021-08-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: High Grade Glioma; Glioblastoma Multiforme
Keywords: High grade glioma; Glioblastoma Multiforme (GMB); Brain Tumor; Emopamil binding protein; 3-beta-hydroxysteroid-Delta(8),Delta(7)-isomerase
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 dose-escalation study with a Part 2 expansion to evaluate the safety, PK, PD, and preliminary antitumor activity of orally administered DSP 0390 in patients with recurrent high-grade glioma. Patients in this study will receive DSP-0390 orally once daily. The study will be divided into 28-day cycles for safety and response assessments. Patients will continue treatment until progression of disease, unacceptable toxicity, withdrawal of consent, loss to follow-up, or discontinuation of the patient by the investigator.
  Dose-escalation will evaluate increasing dose levels of DSP-0390 to determine the MTD and/or a suitable lower dose for expansion (the RDE) in patients with recurrent WHO Grade III or IV malignant glioma. Once the MTD and/or RDE has been established, the dose escalation (Part 2) will evaluate preliminary clinical activity and the safety and tolerability of DSP-0390 in patients with recurrent WHO Grade 4 glioblastoma multiforme (GBM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm DSP-0390 (Experimental): Arm Description [*] DSP-0390 by oral administration
  Interventions: Drug: DSP-0390

INTERVENTIONS:
Drug: DSP-0390 — DSP-0390 administered orally

SUMMARY:
This is a study of DSP-0390 in patients with recurrent high grade glioma.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of DSP-0390 in patients with recurrent high grade glioma.

ELIGIBILITY:
Inclusion Criteria:

Estimated life expectancy >+3 months Recovery from toxic effects of prior therapy to NCI CTCAE v5.0 Grade 1 (non-hematologic toxicities) or Grade <=2(hematologic toxicities, except deep vein thrombosis) KPS >=70%

Adequate organ function as determined by:

* Absolute Neutrophil ≥1500/microliter (may not use G-CSF or GM CSF)
* Platelet ≥100 × 103/microliter
* Hemoglobin ≥9 g/dL (may not transfuse or use erythropoietin to obtain this Hgb level)
* Creatinine Clearance ≥ 40ml/min (Cockcroft-Gault)
* Total bilirubin ≤1.5 times ULN (or ≤ 2 times ULN for patients with known Gilbert's syndrome)
* AST ≤ 3 times ULN
* ALT ≤ 3 times ULN
* INR, PT, PTT, or aPTT ≤1.5 x ULN Note: The use of anticoagulants is permitted as long as the PT/(a)PTT is within therapeutic limits (according to the local institution standard) and the patient has been on a stable anticoagulant regimen for at least 2 weeks prior to study Day 1.

If on antiepileptic drug; dose must be stable and no seizures 14 days prior to study Day 1 If on corticosteroids at baseline, dose must be stable or decreasing for at least 5 days prior to study Day 1. For the dose expansion part of the study, the dose must be ≤ 4 mg dexamethasone per day (or equivalent dose if other corticosteroids are used). A higher stable dose of corticosteroids, if used as HRT, may be allowed upon discussion with the Medical Monitor.

Females of childbearing potential must have a negative serum or urine pregnancy test Male or female patients of child-producing potential must agree to use contraception or use prevention of pregnancy measures or agreement to refrain completely from heterosexual intercourse during the study and for 6 months (females & males) after the last dose of study drug

Exclusion Criteria:

Prior therapy with bevacizumab or other anti-vascular endothelial growth factor (VEGF) treatments within 3 months prior to study Day 1, Multifocal disease, leptomeningeal metastasis, or extracranial metastasis Abnormal ECGs that are clinically significant, including those where QT prolongation (QTcF>450 msec for males and >470 msec for females); and/or history of Torsade de Pointes Left ventricular ejection fraction <40% as determined by ECHO or MUGA Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally Know active Crohn's or other inflammatory bowel disease History of another primary cancer within the 2 years prior to study Day 1, except for the following: non-melamona skin cancer, cervical carcinoma in situ, superficial bladder cancer that has been removed or curatively treated.

Have a known detectable viral load for HIV or HVC, or evidence of a HBV surface antigen, all being indicative of active infection. [Note: Female breastfeeding patients may be enrolled if they interrupt breastfeeding. Breastfeeding should not be resumed for at least 6 months after the last dose of study drug.]

The presence of any active retinal abnormality determined by screening tests using visual acuity, visual field, fundoscopy, and OCT

Significant cardiovascular disease, including NYHA Class III or IV congestive heart failure, myocardial infarction, unstable angina, poorly controlled cardiac arrhythmias, or stroke in the preceding 6 months prior to study Day 1

Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state

Major surgical procedure, surgical resection, open biopsy, or significant traumatic injury within 4 weeks prior to study Day 1 or anticipation of need for major surgical procedure during the course of the study

Minor surgical procedures, fine needle aspirations, or core biopsies within 7 days prior to study Day 1

Evidence of CNS hemorrhage on baseline MRI or CT scan (except for postsurgical, asymptomatic, Gr 1 hemorrhage that has been stable at least 4 weeks for enrolled patients) Chemotherapy or investigational anticancer therapy administered within 4 weeks (except 6 weeks for nitrosoureas and immunotherapy, or 8 weeks for an implanted nitrosoureas wafer) prior to study Day 1

Radiotherapy within 12 weeks prior to study Day 1, unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are 2 MRIs (performed 8 weeks apart) confirming progressive disease

Concurrent use of prohibited medications: carbamazepine, phenytoin, phenobarbital, and other strong or moderate CYP3A4 inhibitors or inducers, and strong CYP2D6 inhibitors. These should be discontinued 1 week or 5 half-lives (whichever is greater) prior to study Day 1

Concurrent treatment with Tumor Treatment Field (Optune) is not allowed. Patients must stop Optune 1 day prior to the first dose of study drug. Any wounds from Optune must be healed adequately prior to study Day 1

History of, within 6 months of study Day 1:

1. Pneumonitis or interstitial lung disease
2. Any other lung condition that in the investigators' judgement may put the patient at an increased risk for lung toxicity (including, but not limited to, suspected interstitial lung disease or radiation-induced lung injury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Assess safety of DSP-0390 by Incidence of TEAEs and SAEs in adult patients with recurrent high-grade glioma | From date of treatment through 30 days after End of Treatment an average of 6 months
  Occurrence of DLTs by Incidence of TEAEs and SAEs, as assessed by NCI CTCAE v5.0
Dose Escalation: Assess safety of DSP-0390 by severity of TEAEs and SAEs in adult patients with recurrent high-grade glioma | From date of treatment through 30 days after End of Treatment an average of 6 months
  Occurrence of DLTs by severity of TEAEs and SAEs, as assessed by NCI CTCAE v5.0
Dose Escalation: Determine the MTD and/or RDE of DSP-0390 | From date of first treatment through Cycle 1 (28-day cycle) DLT monitoring period
  Incidence of dose-limiting toxicities
Dose Expansion: Evaluate the change in Baseline tumor activity of DSP-0390 using radiologic assessments. | From date of first treatment, assessed by radiologic examination performed at 8-week intervals through study completion, an average of 6 months
  Evaluate the change in baseline tumor activity of DSP-0390 using radiologic assessments evaluated by RANO 2010 Evaluation Criteria
Dose Expansion: Evaluate the safety of the Recommended Phase 2 Dose of DSP-0390 by assessment of incidence of TEAEs and SAEs | From date of first treatment through study completion, an average of 6 months
  Assess the safety of the Recommended Phase 2 Dose of DSP-0390 by assessment of incidence of TEAEs and SAEs
Dose Expansion: Evaluate the safety of the Recommended Phase 2 Dose by assessment of severity of TEAEs and SAEs | From date of first treatment through study completion, an average of 6 months
  Assess the safety of the Recommended Phase 2 Dose of DSP-0390 by assessment of severity of TEAEs and SAEs
Assess safety of DSP-0390 by Incidence of SAEs in adult patients with recurrent high-grade glioma consented under Protocol Amendment 5 | From date of treatment through 30 days after End of Treatment an average of 12 months
  Incidence of SAEs, as assessed by NCI CTCAE v5.0
Assess safety of DSP-0390 by Incidence of AEs resulting in study discontinuation in adult patients with recurrent high-grade glioma consented under Protocol Amendment 5 | From date of treatment through 30 days after End of Treatment an average of 12 months
  Incidence of AEs resulting in study discontinuation, as assessed by NCI CTCAE v5.0

SECONDARY OUTCOMES:
Dose Escalation: Characterize the PK profile for AUC | Cycle 1 Day 1 and Cycle 2 Day 1- 0, 30 min, and 1, 2, 4, 6, 8, 10, 12 hrs, each cycle is 28 days
  PK assessed for AUC
Dose Escalation: Characterize the PK profile for Cmax | Cycle 1 Day 1 and Cycle 2 Day 1 -0, 30 min, and 1, 2, 4, 6, 8, 10, 12 hrs , each cycle is 28 days
  PK assessed for Cmax
Dose Escalation: Characterize the PK profile for tmax | Cycle 1 Day 1 and Cycle 2 Day 1- 0, 30 min, and 1, 2, 4, 6, 8, 10, 12 hrs , each cycle is 28 days
  PK assessed for tmax
Dose Escalation: Characterize the PK profile for t1/2 | From date of first treatment, Cycle 1 Day 1 and Cycle 2 Day 1- 0, 30 min, and 1, 2, 4, 6, 8, 10, 12 hrs , each cycle is 28 days]
  PK assessed for t1/2
Dose Escalation: Characterize the PK profile for Racc | Cycle 1 Day 8, 15 and 22 and Cycle 2 Day 1, each cycle is 28 days
  PK assessed for Racc
Dose Escalation: Evaluate preliminary antitumor activity | From date of first treatment, assessed by radiologic examination performed at 8-week intervals through study completion, an average of 6 months]
  Objective response (complete or partial response) and duration of response assessed by RANO criteria.

OTHER OUTCOMES:
Exploratory: Assess the PD effect of DSP-0390 | From first date of treatment, blood tests performed at 8 week intervals through study completion, an average of 6 months
  Biomarker (lathosterol/zymostenol ratio) in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (9):
- United States (6):
  - University of California at San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Japan (3):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyoto University Hospital, Kyoto, Sakyo-ku
  - National Cancer Center Hospital, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No